CLINICAL TRIAL: NCT00746382
Title: A Proof of Concept Study With 0.5% Roflumilast Cream in Patients With Mild Atopic Dermatitis
Brief Title: A Placebo Controlled 4 Week Proof of Concept Study With 0.5% Roflumilast Cream in Patients With Mild Atopic Dermatitis (RO-2351-001-EM)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to business decisions. No subjects were treated.
Sponsor: AstraZeneca (Industry)
Collaborators: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO-2351-001-EM
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Dermatitis
Keywords: Mild atopic dermatitis, Roflumilast cream 0.5%
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Roflumilast cream 0.5%
  Interventions: Drug: Roflumilast cream
- 2 (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Roflumilast cream — Roflumilast cream 0.5% versus Placebo cream
  Arms: 1
Drug: Placebo cream — Placebo cream
  Arms: 2

SUMMARY:
The aim of this proof of concept study is to show the safety and efficacy of 0.5 % dermal roflumilast cream in the treatment of atopic dermatitis in adults. This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study. 2-5 % of the body surface area (BSA) should be covered with a mild form of atopic dermatitis. In a 4-week treatment period 38 mg cream is applied two times daily on 0.5 to 1 % of the BSA. After a screening phase, a washout phase of flexible duration (max 30 days, time depending upon pre-medication), the 28 day treatment phase follows.As roflumilast is a potent antiinflammatory substance, a positive effect on this form of dermal disease is anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Patient /who is able to read, to write and to fully understand English language) has been informed both verbally and in writing about the objectives of the clinical study, the methods, the anticipated benefits and potential risks and the discomfort to which he/she may be exposed, and has given written consent to participation in the study prior to study start and any study-related procedure.
* Patients are suffering from mild, stable atopic dermatitis Male or female patient of any ethnic origin, age 18 years or older presenting a minimum of 2% to a maximum of 5% BSA affected by stable mild atopic dermatitis (IgE > 10)proven by a dermatologist.
* Patients must have at least one target lesion of at least 0.5% BSA.
* No evidence of oozing or crusting atopic dermatitis
* No lichenification of diseased lesions
* No excoriation of diseased lesions
* Patients must be willing to wash out from current active therapy for at least 14 days to Day 1.
* Women of childbearing potential must have a negative pregnancy test at the Screening and Baseline Visits and agree to use a highly effective method of birth control. A highly effective of birth control is defined at those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectable, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.

Exclusion Criteria:

* Patient has spontaneously improving or rapidly deteriorating atopic dermatitis.
* Patient has a physical condition which, in the Investigator´s opinion, might impair evaluation of atopic dermatitis or which exposes the patient to an unacceptable risk by study participation.
* Patient had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to the initiation of treatment or is intending to have such exposure during the study that is thought by the Investigator likely to modify the patient´s disease.
* The patient had topical or transdermal treatments, such as but not limited to retinoids, nicotine or hormone replacement therapies, on or near the intended site of application within 14 days prior to first application of study medication. Use of other topical preparations such as those containing vitamins, supplements or herbal within 14 days prior to application.
* Treatment with systemic/locally acting medications/procedures which might counter or influence the study aim within 30 days before the start and during the study /e.g. anti-histamines, topical glucocorticosteroids, pimecrolimus , tacrolimus systematic desensitization)
* Patient is pregnant, nursing or planning a pregnancy during the study period.
* Patient has received an investigational drug or an investigational device within 30 days prior to study start.
* Abuse of alcohol or drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of clinical signs and symptoms score, improvement of patient judged pruritus severity | 28 days

SECONDARY OUTCOMES:
Improvement of atopic dermatitis severity score, change in dermal questionaire, safety and efficacy | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca